CLINICAL TRIAL: NCT04187586
Title: Effect of Extracorporeal Shock Wave Therapy for Burn Scar Charateristics: A Retrospective Study
Brief Title: Effect of Extracorporeal Shock Wave Therapy for Burn Scar Charateristics
Status: Completed | Type: Observational
Sponsor: Hangang Sacred Heart Hospital (Other)
Collaborators: Hallym University (Other)
Responsible Party: Sponsor
Other Study IDs: HangangSHH-9
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-12

CONDITIONS: Burn Scar
Keywords: burns; rehabilitation; extracorporeal shock wave therapy
MeSH Terms: conditions — Burns | interventions — Extracorporeal Shockwave Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Extracorporeal shock wave therapy group: The ESWT group received shock waves with low-energy flux density (0.05-0.30 mJ/mm2). The interval between treatments is a 1-week. To evaluate the effect of ESWT, we reviewed the skin test results (thickness, melanin, erythema, TEWL, sebum, and skin elasticity levels) immediately before ESWT and immediately after the sixth session. And also the ESWT group received the standard treatment, which involved medication, scar lubrication, burn rehabilitation massage therapy, and physical therapy.
  Interventions: Other: Extracorporeal shock wave therapy
- conventional therapy without extracorporeal shock wave therapy: Conventional therapy group received the standard treatment, which involved medication, scar lubrication, burn rehabilitation massage therapy, and physical therapy.

INTERVENTIONS:
Other: Extracorporeal shock wave therapy — ESWT was performed around the primary treatment site at 100 impulses/cm2, an energy flux density(EFD) of 0.05 to 0.30 mJ/mm2, frequency of 4Hz, and 1000 to 2000 impulses were administered at 1-week intervals for 6 sessions.
  Groups: Extracorporeal shock wave therapy group

SUMMARY:
No study has investigated the effect of extracorporeal shock wave therapy (ESWT) on hypertrophic scar characteristics. Thus, this study aimed to ascertain the effects ESWT on burn scars. The investigators retrospectively reviewed burn patients who had undergone autologous split-thickness skin grafting (STSG) with same artificial dermis between January 2012 and September 2019.

DETAILED DESCRIPTION:
No study has investigated the effect of extracorporeal shock wave therapy (ESWT) on hypertrophic scar characteristics. Thus, this study aimed to ascertain the effects ESWT on burn scars. The investigators retrospectively reviewed burn patients who had undergone autologous split-thickness skin grafting (STSG) with same artificial dermis between January 2012 and September 2019. The ESWT group (n=17) received shock waves with low-energy flux density (0.05-0.30 mJ/mm2). The interval between treatments is a 1-week. The ESWT group also received standard treatment. The control group (n=18) only received standard treatment. We reviewed skin characteristics before and after 6 treatment sessions for both groups. The investigators checked skin charateristics(erythema, transepidermal water loss, sebum level, and elasticity). The investigators expect that ESWT is effective for significantly improving burn-associated scar characteristics and may be used for managing burn patients.

ELIGIBILITY:
Inclusion Criteria:

* a retrospective review of 35 patients who had undergone STSG between January 2012 and September 2019
* limited to the upper extremities(the upper arm, forearm, and hand)
* the scars which undergone STSG with same artificial dermis using Matriderm® (MeSkin Solution Dr. Suwelack AG, Billerbeck, Germany)

Exclusion Criteria:

* not evaluated serial assessments
* below 18 years age

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: * This study was a retrospective review of 35 patients who had undergone STSG using Matriderm® (MeSkin Solution Dr. Suwelack AG, Billerbeck, Germany) between January 2012 and September 2019.
  * The subjects who were admitted to the Department of Rehabilitation Medicine at Hangang Sacred Heart Hospital were enrolled.
Sampling Method: Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
scar thickness | 6 weeks
  hypertrophic scar thickness check using ultrasonic wave equipment (128 BW1 Medison, Korea).

SECONDARY OUTCOMES:
scar erythema | 6 weeks
  pigementation and erythema check using Mexameter® (MX18, Courage-Khazaka Electronics GmbH, Germany). The higher values indicating a darker and redder skin.
scar transepidermal water loss(TEWL) | 6 weeks
  TEWL measured with a Tewameter® (Courage-Khazaka Electronic GmbH, Germany), which is used for evaluating water evaporation. The higher values indicating a skin dryness.
Sebum | 6 weeks
  Sebum in the scars was measured with the Sebumeter® (Courage-Khazaka Electronic GmbH, Germany). The measurement is based on the principle of grease-spot photometry using a cassette with its special tape. A microprocessor calculates the result, which is shown on the display in mg/cm2.
Elasticity | 6 weeks
  Elasticity was measured using Cutometer SEM 580® (Courage-Khazaka Electronic GmbH, Cologne, Germany), which applies negative pressure (450 mbar) on the skin. The numeric values (mm) of the skin's distortion is presented as the elasticity. Two seconds of negative pressure of 450 mbar is followed by 2 s of recess, and this consists of a complete cycle. Three measurement cycles were conducted, and the average values were obtained. The higher values present the higher elasticity.

CONTACTS AND LOCATIONS:
Locations (1):
- Hangang Sacred Heart Hospital, Seoul, Yeong-deungpo-Dong, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cui HS, Hong AR, Kim JB, Yu JH, Cho YS, Joo SY, Seo CH. Extracorporeal Shock Wave Therapy Alters the Expression of Fibrosis-Related Molecules in Fibroblast Derived from Human Hypertrophic Scar. Int J Mol Sci. 2018 Jan 2;19(1):124. doi: 10.3390/ijms19010124. PMID 29301325
- [Background] Joo SY, Cho YS, Seo CH. The clinical utility of extracorporeal shock wave therapy for burn pruritus: A prospective, randomized, single-blind study. Burns. 2018 May;44(3):612-619. doi: 10.1016/j.burns.2017.09.014. Epub 2017 Oct 10. PMID 29029857
- [Background] Cho YS, Joo SY, Cui H, Cho SR, Yim H, Seo CH. Effect of extracorporeal shock wave therapy on scar pain in burn patients: A prospective, randomized, single-blind, placebo-controlled study. Medicine (Baltimore). 2016 Aug;95(32):e4575. doi: 10.1097/MD.0000000000004575. PMID 27512886